CLINICAL TRIAL: NCT00002892
Title: A RANDOMISED STUDY OF OBSERVATION VERSUS ADJUVANT LOW DOSE EXTENDED DURATION INTERFERON ALPHA-2A IN COMPLETELY RESECTED HIGH RISK MALIGNANT MELANOMA
Brief Title: Interferon Alfa or No Further Therapy Following Surgery in Treating Patients With Stage II, Stage III, or Recurrent Melanoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065215; NCRI-AIM-HIGH; EU-96052; UKCCCR-AIM-HIGH
Record Dates: First submitted 1999-11-01; First posted 2004-05-13 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2007-05

CONDITIONS: Melanoma (Skin)
Keywords: stage II melanoma; stage III melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Interferon-alpha

INTERVENTIONS:
Biological: recombinant interferon alfa

SUMMARY:
RATIONALE: Interferon alfa may interfere with the growth of the cancer cells. It is not yet known whether interferon alfa following surgery is more effective than surgery alone in treating patients with melanoma.

PURPOSE: Randomized phase III trial to compare the effectiveness of interferon alfa with no further therapy following surgery in treating patients with stage II, stage III, or recurrent melanoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the effects of adjuvant low-dose extended-duration interferon alfa on disease-free and overall survival in patients with completely resected malignant melanoma at high risk of recurrence. II. Determine any correlation between patient age or sex and the effects of interferon therapy on disease-free and overall survival. III. Describe the toxic effects of this treatment. IV. Evaluate the economic implications of implementing effective interferon therapy in these patients.

OUTLINE: This is a randomized study. Patients will be stratified by age, sex, disease status at entry, and participating institution. Patients are randomized to observation only or to receive interferon alfa by subcutaneous injections 3 times weekly for 2 years, or until disease progression or toxicity intervenes. Patients are followed monthly for 6 months, quarterly for 18 months, and every 6 months thereafter.

PROJECTED ACCRUAL: A total of 1,000 patients will be entered over 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed malignant melanoma definitively resected within 12 weeks prior to entry One of the following categories: Stage II disease (greater than 4 mm Breslow thickness) Stage III disease (regional lymph node involvement) Recurrent non-nodal superficial regional disease (local or in transit) Recurrent regional nodal involvement

PATIENT CHARACTERISTICS: Able to tolerate interferon No second malignancy except curatively treated: Carcinoma of the cervix Nonmelanomatous skin cancer No pregnant or nursing women

PRIOR CONCURRENT THERAPY: No prior immunosuppressive therapy, including systemic steroids No prior biologic therapy Recovered from surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 1995-10; Study Completion 2001-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry W. Hancock, MD, Study Chair — Cancer Research Centre at Weston Park Hospital
Locations (14):
- United Kingdom (14):
  - Royal Free Hospital, Hampstead, London, England
  - St. James's Hospital, Leeds, England
  - University Hospitals of Leicester, Leicester, England
  - Guy's, King's and St. Thomas' Hospitals Trust, London, England
  - Royal Marsden NHS Trust, London, England
  - Christie Hospital N.H.S. Trust, Manchester, England
  - Clatterbridge Centre for Oncology NHS Trust, Merseyside, England
  - Weston Park Hospital, Sheffield, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Selly Oak Hospital, Birmingham
  - Royal Bournemouth Hospital, Bournemouth
  - Queen Elizabeth Hospital, Kings Lynn
  - Salisbury District Hospital, Salisbury
  - Southend Hospital, Southend-on-Sea

REFERENCES:
- [Result] Hancock BW, Wheatley K, Harris S, Ives N, Harrison G, Horsman JM, Middleton MR, Thatcher N, Lorigan PC, Marsden JR, Burrows L, Gore M. Adjuvant interferon in high-risk melanoma: the AIM HIGH Study--United Kingdom Coordinating Committee on Cancer Research randomized study of adjuvant low-dose extended-duration interferon Alfa-2a in high-risk resected malignant melanoma. J Clin Oncol. 2004 Jan 1;22(1):53-61. doi: 10.1200/JCO.2004.03.185. Epub 2003 Dec 9. PMID 14665609